CLINICAL TRIAL: NCT00006100
Title: A Phase I Pilot Trial to Evaluate the Toxicity of Epstein-Barr Virus Specific T-Lymphocytes or Peripheral Blood Mononuclear Cells for the Treatment of Relapsed/Refractory Hodgkin's Disease
Brief Title: Allogeneic Epstein Barr Virus-Specific Cytotoxic T-Lymphocytes in Treating Patients With Progressive, Relapsed, or Refractory Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068109; PSCI-2003-257; UAB-0002; NCI-G00-1829
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2005-05

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — aldesleukin; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: aldesleukin
Biological: allogeneic Epstein-Barr virus-specific cytotoxic T lymphocytes
Drug: fludarabine phosphate
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Donor white blood cells that are treated in the laboratory with Epstein-Barr virus may be effective treatment for Hodgkin's lymphoma.

PURPOSE: Phase I trial to study the effectiveness of allogeneic Epstein-Barr virus-specific cytotoxic T cells in treating patients who have progressive, relapsed, or refractory Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of allogeneic Epstein Barr virus (EBV)-specific cytotoxic T-lymphocytes (EBV CTL) in patients with progressive, relapsed, or refractory EBV-positive Hodgkin's lymphoma.
* Detect alterations in the anti-EBV cellular immunity of patients treated with EBV CTL.

OUTLINE: Donors undergo leukapheresis. Epstein Barr virus-specific cytotoxic T lymphocytes (EBV CTL) are cultured in vitro.

Patients receive an infusion of EBV CTL over 10 minutes on day 0. The EBV CTL infusion is preceded by 3 doses of fludarabine. Patients then receive interleukin-2 injections for 12 days after the EBV CTL infusion.

Patients are followed weekly for 1.5 months, twice a month for 1.5 months, and then monthly for 3 months.

PROJECTED ACCRUAL: A total of 9 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven Hodgkin's lymphoma

  * Progressive, relapsed, or refractory disease after prior chemotherapy, radiotherapy, and/or stem cell transplantation
  * Epstein Barr virus (EBV) positive by immunohistochemical staining for LMP-1 or 2 OR the presence of EBV RNA (EBER)
* Availability of an HLA identical or haploidentical donor for cytotoxic T-lymphocytes, meeting the following criteria:

  * EBV seropositive
  * HIV negative
  * HTLV-1 negative
  * Hepatitis B surface antigen and hepatitis B core antibody IgM negative
  * Hepatitis C antibody negative
  * Must share at least 1 HLA haplotype with donor

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* Not specified

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGOT/SGPT less than 2.5 times normal (unless liver metastases are present)

  * If there is liver involvement by disease, an obvious relationship between SGOT/SGPT and disease activity is required
* No hepatic dysfunction causing moribundity

Renal:

* Creatinine clearance greater than 50 mL/min
* No renal dysfunction causing moribundity

Cardiovascular:

* No cardiac dysfunction causing moribundity

Pulmonary:

* No pulmonary dysfunction causing moribundity

Other:

* No neurologic dysfunction causing moribundity
* No history of severe transfusion reactions with blood products (including fetal calf serum)
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics
* No concurrent antimetabolites

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-04

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G. Lucas, MD, Study Chair — Milton S. Hershey Medical Center
Locations (1):
- Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Result] Lucas KG, Salzman D, Garcia A, Sun Q. Adoptive immunotherapy with allogeneic Epstein-Barr virus (EBV)-specific cytotoxic T-lymphocytes for recurrent, EBV-positive Hodgkin disease. Cancer. 2004 May 1;100(9):1892-901. doi: 10.1002/cncr.20188. PMID 15112270